CLINICAL TRIAL: NCT03915626
Title: Determination of Serum Rivastigmine Levels After Using Rivastigmine Transdermal Delivery Systems With and Without Standardized Heat Application in Healthy Human Volunteers
Brief Title: Effect of Heat on Rivastigmine TDS Products
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Audra Stinchcomb, Professor, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HP-00076010
Record Dates: First submitted 2019-03-05; First posted 2019-04-16 (Actual); Results first posted 2022-03-07 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Bioavailability
MeSH Terms: interventions — Rivastigmine; Transdermal Patch; Drugs, Generic

STUDY DESIGN:
Intervention Model Description: The same healthy subjects are assigned to all four treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- RLD patch (Experimental): RLD rivastigmine patch (4.6 mg/24 hours); worn for 9 hours
  Interventions: Drug: Rivastigmine (RLD) transdermal patch
- generic patch (Experimental): generic rivastigmine patch (4.6 mg/24 hours); worn for 9 hours
  Interventions: Drug: Rivastigmine (generic) transdermal patch
- RLD patch with heat (Experimental): RLD rivastigmine patch (4.6 mg/24 hours); worn for 9 hours; 90 min heat application
  Interventions: Drug: Rivastigmine (RLD) transdermal patch
- generic patch with heat (Experimental): generic rivastigmine patch (4.6 mg/24 hours); worn for 9 hours; 90 min heat application
  Interventions: Drug: Rivastigmine (generic) transdermal patch

INTERVENTIONS:
Drug: Rivastigmine (RLD) transdermal patch — brand name patch
  Other Names: brand name patch
  Arms: RLD patch; RLD patch with heat
Drug: Rivastigmine (generic) transdermal patch — generic patch
  Other Names: generic patch
  Arms: generic patch; generic patch with heat

SUMMARY:
This research study is designed to measure the amount of medicine in blood over time after the patch is placed on the skin with and without external heat application.

ELIGIBILITY:
Inclusion Criteria:

1. Men or non-pregnant, non-lactating women who are of any ethnic background between the age of 18 to 45 years old
2. Subjects must be non-smokers/tobacco users (must have refrained from the use of nicotine-containing substances, including tobacco products (e.g., cigarettes, cigars, chewing tobacco, snuff, gum, patches or electronic cigarettes) over the previous 2 months and are not currently using tobacco products
3. Provide written informed consent before initiation of any of the study procedures
4. Agree not to participate in another clinical trial/study or to participate in an investigational drug study for at least one month after the last study session
5. Able to adhere to the study restrictions and protocol schedule
6. Able to participate in all study sessions
7. Subjects deemed to be healthy as judged by the Medically Accountable Investigator (MAI) and determined by medical history, physical examination and medication history
8. Negative urine drug screening test (cannabinoids, amphetamines, barbiturates, benzodiazepine, cocaine, methadone, opiates, PCP)
9. Have normal screening laboratories for white blood cells (WBC), hemoglobin (Hgb), platelets, sodium, potassium, chloride, bicarbonate, blood urea nitrogen (BUN), creatinine, alanine transaminase (ALT) and aspartate aminotransferase (AST)
10. Have normal screening laboratories for urine protein and urine glucose
11. Female subjects must be of non-childbearing potential (as defined as surgically sterile [i.e. history of hysterectomy or tubal ligation] or postmenopausal for more than 1 year), or if of childbearing potential must be non-pregnant at the time of enrollment and on the morning of each procedure day, and must agree to use reliable hormonal or barrier birth control such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or a vasectomized partner
12. Agree not to donate blood to a blood bank throughout participation in the study and for at least three months after last procedure day
13. Have a normal ECG; must not have the following to be acceptable: pathologic Q wave abnormalities, significant ST-T wave changes, left ventricular hypertrophy, right bundle branch block, left bundle branch block. (sinus rhythm is between 55-100 beats per minute)
14. Have normal vital signs:

    * Temperature 35-37.9°C (95-100.3°F)
    * Systolic blood pressure 90-140 mmHg
    * Diastolic blood pressure 60-90 mmHg
    * Heart rate 55-100 beats per minute
    * Respiration rate 12-20 breaths per minute

Exclusion Criteria:

1. Women who are pregnant, lactating, breast feeding or have a positive serum pregnancy test at enrollment or positive urine pregnancy test on the morning of any study session
2. Smokers/tobacco users (current use or use over the previous 2 months of nicotine-containing substances, including tobacco products (e.g., cigarettes, cigars, chewing tobacco, snuff, gum, patch or electronic cigarettes)
3. Participation in any ongoing investigational drug trial/study or clinical drug trial/study
4. History of lung, heart, respiratory or blood disease
5. Active positive Hepatitis B, C and/or HIV serologies
6. Positive urine drug screening test
7. Use of chronic prescription medications during the period 0 to 30 days; or over-the-counter medications (e.g. cholinomimetic drugs [used to treat diseases like acid reflux in children, glaucoma, dry mouth associated with Sjögren's Syndrome], anticholinergics [used to treat diseases like asthma, incontinence, gastrointestinal cramps, and muscular spasms], antihistamines, topical corticosteroids) and short term (<30 days) prescription medications during the period 0-3 days before a study session vitamin, herbal supplements and birth control medications not included)
8. Donation or loss of greater than one pint of blood within 60 days of entry to the study
9. Any prior allergies to rivastigmine, other carbamate derivatives, other ingredients in the patch, to medical tape products or other skin patches
10. Subject has problems with urinary retention, gastric retention or gastrointestinal obstruction
11. Subject has continuous spasms, muscle contractions, motor restlessness, rigidity, slowness of movement, tremors or irregular jerky movements
12. Subject has ulcers or gastrointestinal bleeding
13. Subject has asthma or blocked airflow making it hard to breathe (COPD)
14. Received an experimental agent (vaccine, drug, biologic, device, blood product or medication) within one month before enrollment in this study or expects to receive an experimental agent during the study
15. Any condition that would, in the opinion of the Medically Accountable Investigator (MAI), place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol
16. Consumption (food or drink) of alcohol within 24 h prior to dose administration
17. History as either reported by the subject or evident to the investigator of infectious disease or skin infection or of chronic skin disease (e.g., psoriasis, atopic dermatitis)
18. History of diabetes
19. Hereditary skin disorders or any skin inflammatory conditions as reported by the subject or evident to the MAI
20. History of significant dermatologic cancers (e.g., melanoma, squamous cell carcinoma) except basal cell carcinomas that were superficial and did not involve the investigative sites
21. Subject has an obvious difference in skin color between arms or the presence of a skin condition, excessive hair at the application site (upper arms), sunburn, raised moles and scars, open sores at application site (upper arms), scar tissue, tattoo, or coloration that would interfere with placement of products, skin assessment, or reactions to rivastigmine
22. BMI ≥30 kg/m2

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Audra L Stinchcomb, PhD, Principal Investigator — University of Maryland, Baltimore School of Pharmacy
Locations (1):
- General Clinical Research Center (GCRC) at the University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Rivastigmine RLD and Generic Patches: Session 1: RLD patch worn for 9 hours, then at least one week wash out period, Session 2: Generic patch worn for 9 hours, then at least one week wash out period, Session 3: RLD patch worn for 9 hours includes 90 minute heat application (5 h-6 h 30 min), then at least one week wash out period Session 4: Generic patch worn for 9 hours includes 90 minute heat application (5 h-6 h 30 min)
Period: Overall Study
Arm/Group | Rivastigmine RLD and Generic Patches
Started (Study was intended to enroll and complete n=12 volunteers; however, funding was terminated due to pandemic.) | 7
Completed | 6
Not Completed | 1
Not completed — study was halted due to COVID-19; once started again volunteer could no longer participate | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rivastigmine RLD and Generic Patches
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.57 (4.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Total Area Under the Curve (AUC) 0-12 Hours
Description: Blood samples were obtained at the following time points: -60 min (before patch application) and then 2 h, 3 h, 4 h, 5 h, 5 h 15 min, 5 h 30 min, 5 h 45 min, 6 h, 6 h 15 min, 6 h 30 min, 6 h 45 min, 7 h, 7 h 30 min, 8 h, 8 h 30 min, 9 h, 9 h 15 min, 9 h 30 min, 10 h, 11 h, 12 h post patch administration.
Time Frame: 0-12 hours for each subject for each of the four study sessions
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | RLD Patch | Generic Patch | RLD Patch With Heat | Generic Patch With Heat
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng*h/mL | 19.99 (14.35) | 19.22 (11.41) | 19.22 (11.41) | 16.57 (9.66)

ADVERSE EVENTS:
Time Frame: Subjects were observed for the 12 hours during product administration and then were followed up with a phone call up to 72 h after product removal; ~4 days for each of the four study sessions.
Arm/Group | RLD Patch | Generic Patch | RLD Patch With Heat | Generic Patch With Heat
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7 | 4/6 | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RLD Patch (N=7) | Generic Patch (N=7) | RLD Patch With Heat (N=6) | Generic Patch With Heat (N=6)
Dizziness (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased heart rate (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased heart rate (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased blood pressure (Cardiac disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Increased blood pressure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
SOMNOLENCE (SLEEPINESS) (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ERYTHEMA (skin reddening) (Skin and subcutaneous tissue disorders) | 7 (7) | 7 (7) | 4 (6) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT03915626/Prot_SAP_000.pdf